CLINICAL TRIAL: NCT01576237
Title: Open Prospective Multi-national Long-term Study to Register Adverse Events Related to Hemaphereses by Means of an Internet-based Haemapheresis Vigilance Questionnaire
Brief Title: Multinational Haemapheresis Vigilance Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: DGTI - Haemapheresis Vigilance Working Party (Network)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Other Study IDs: DGTI-AGHV_01
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Blood Donation With Hemapheresis
Keywords: hemovigilance; hemapheresis; donor vigilance; plasmapheresis; platelet apheresis; leukapheresis; stem cell apheresis; granulocyte apheresis; monocyte apheresis; red cell apheresis
MeSH Terms: interventions — Blood Donation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy apheresis donors: healthy blood donors for blood cell aphereses
  Interventions: Other: blood donation

INTERVENTIONS:
Other: blood donation — blood donation with preparative hemapheresis

SUMMARY:
During a seven years period the participating transfusion medicine establishments will report all their non-trivial adverse events (AE) occurring during preparative hemaphereses. Complications may be related to the blood donors, the blood products, the disposables or the apheresis devices. The study hypothesis regarding each participating center is that their procedure-related AE rate is not higher than the respective rate of all other centers in total.

DETAILED DESCRIPTION:
In the scope of this study the participating transfusion medicine establishments obligate themselves to record all significant Adverse Events (AE) related to preparative hemaphereses of healthy donors. All complications (phlebotomy and circulation problems, citrate toxicity, donor compliance, and technical complications) shall be assessed with respect to plasma-, platelet-, leukocyte- (stem cells, granulocytes, monocytes), and red cell aphereses as well as multicomponent aphereses. Study data are recorded by means of an Internet-based hemapheresis vigilance system. Study results will be evaluated according to the advanced standards of the International Haemovigilance Network (IHN). The study contributes to the quality assurance of each single center as it enables the comparison to other transfusion medicine establishments.

ELIGIBILITY:
Inclusion Criteria:

* blood donor standard criteria :
* healthy donor of > 50 kg
* hemoglobin 125 g/L or 7.8 mmol/L (female donors)
* hemoglobin 135 g/L or 8.4 mmol/L (male donors)
* hemoglobin > 140 g/L for 2 unit red cell apheresis
* total proteins >= 60 g/L for plasmapheresis
* platelet count >= 150 × 10e9/L for platelet apheresis
* blood volume of > 5 L for 2 unit red cell apheresis
* normal leukocyte count

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all blood donors having an Adverse Event during preparative cell aphereses
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of all non-trivial adverse events (AE) occurring during hemapheresis | up to one year
  All non-trivial AEs will be recorded regardless of whether anticipated products have been collected or not

SECONDARY OUTCOMES:
Rate of products per apheresis | hemapheresis stay: expected time range from 1 hour for plasmaphereses to 5 hours for stem cell aphereses
  amount of obtained products vs. anticipated products

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Gert Heuft, PD. Dr. med., Principal Investigator — Hannover Medical School (MHH)

REFERENCES:
- See also: European Donor Haemovigilance system (EDoH) — http://haemovigilance.eu/
- See also: European Donor Haemovigilance system (EDoH) — http://haemovigilance.com